CLINICAL TRIAL: NCT05202756
Title: Examining Feasibility, Acceptability, and Sustainability of a Novel Personalized Smartphone Intervention for Suicide
Brief Title: Examining Feasibility, Acceptability, and Sustainability of a Novel Personalized Smartphone Intervention for Suicide - Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1678556; R34MH124971 (NIH)
Record Dates: First submitted 2022-01-03; First posted 2022-01-21 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Suicide and Self-harm; Suicide; Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide; Self-Injurious Behavior; Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application to Prevent Suicide (MAPS) (Experimental): Participants receiving MAPS will receive the Safety Planning Intervention (SPI) which will be uploaded into the smartphone app. They will be prompted four times per day to complete a brief ecological momentary assessment "check-in" inquiring about their cognitions, affect, and behavior, including suicidal thoughts and behaviors. Based on these responses, they will be provided with coping strategies from their safety plans and from a database of coping strategies created by study staff. They will also have access to emergency phone numbers, the coping strategies database, and can communicate with their study clinician through a text-like interface in the app. They will receive this intervention for one month.
  Interventions: Behavioral: Mobile Application to Prevent Suicide (MAPS)
- EMA Monitoring Only (EMO) (Active Comparator): Participants in this condition will receive the Safety Planning Intervention (SPI) and will receive ecological momentary assessment prompts on the same schedule as the MAPS condition. However, they will not have access to any other MAPS features.
  Interventions: Behavioral: EMA Monitoring Only

INTERVENTIONS:
Behavioral: Mobile Application to Prevent Suicide (MAPS) — Safety Planning Intervention, ecological momentary intervention smartphone app system, and bidirectional communication with study clinician.
  Arms: Mobile Application to Prevent Suicide (MAPS)
Behavioral: EMA Monitoring Only — Safety Planning Intervention; ecological momentary assessment only
  Arms: EMA Monitoring Only (EMO)

SUMMARY:
The primary aim of the present study is leverage existing infrastructure to develop novel technological features for a novel personalized smartphone intervention system, called the Mobile Application to Prevent Suicide (MAPS), and to establish feasibility, acceptability, safety, and estimate key parameters for primary outcomes (i.e., suicidal ideation and behavior; re-hospitalization), and target mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Presence of suicidal ideation and/or suicidal behavior in the past month
* Between the ages of 18 and 70
* Able to read, write, and understand English well enough to complete study procedures
* Owns a smartphone

Exclusion Criteria:

* Current psychotic or manic symptoms severe enough to interfere with completion of study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 1 month
  Measured using the Client Satisfaction Questionnaire, a self-report measure of satisfaction with treatment. Scores range from 8 to 32, with higher scores representing higher satisfaction.
Acceptability of Research (Recruitment) | Baseline
  Measured by recruitment rate.
Acceptability of Research (Dropout) | 6 months
  Measured by dropout rate.
Acceptability of Research Procedures | 1 month
  Feedback on qualitative interview.
Acceptability of MAPS Intervention | 1 month
  Feedback on qualitative interview.
Satisfaction with MAPS Intervention | 4 weeks
  Measured by protocol completion rate.
Ecological Momentary Assessment (EMA) Adherence | 4 weeks
  Number of assessments completed out of total
Suicidal Ideation and Behavior | 6 months
  Will be assessed using the Columbia Suicide Severity Rating Scale, items from the Modified Scale for Suicidal Ideation, and ecological momentary assessment of suicidal ideation and behavior. The Columbia Suicide Severity Rating Scale can provide presence/absence of suicidal ideation and suicidal behavior, as well as a suicidal ideation score ranging from 0 to 5 with higher scores representing more severe ideation, and a suicidal ideation intensity rating from 0-25 with higher scores representing more intense ideation.
Rehospitalization | 6 months
  Number of inpatient rehospitalizations will be assessed using the Treatment History Interview and medical records review.
Emergency Department Visits | 6 months
  Number of emergency department visits will be assessed using the Treatment History Interview and medical records review.

SECONDARY OUTCOMES:
Use of MAPS Intervention-delivered Coping Strategies (target mechanism) | 4 weeks
  Coping strategy use will be measured in three ways: (1) when participants are prompted to use a coping strategy via MAPS, followup prompts ask whether or not they used the coping skill, (2) in each EMA survey, participants are asked whether or not they used any coping skills since the last survey, and (3) the system provides output with regard to how many times participants dial a support contact phone number through the MAPS app.
Reduction of Negative Affect (target mechanism) | 4 weeks
  Negative affect will be measured using Positive and Negative Affect Scale (PANAS-X) items on ecological momentary assessment surveys. Each emotion item on the PANAS-X is rated on a 1-5 scale based on how participants feel, with 1 indicating "very slightly or not at all" and 5 indicating "extremely."
Self-Efficacy (target mechanism) | 4 weeks
  Coping self-efficacy will be measured using the Coping Self-Efficacy Scale. Self-efficacy for seeking mental health care will be measured by the Self-Efficacy to Seek Mental Health Care Scale. The total score can range from 0-260; the higher the score, the higher the level of coping self-efficacy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Butler Hospital, Providence, Rhode Island
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
After all data have been collected and the results of the studies published, de-identified data will be made available to other qualified researchers on request.